CLINICAL TRIAL: NCT06658457
Title: Investigation of Factors That May Affect Headache in Individuals With Juvenile Onset Systemic Lupus Erythematosus
Brief Title: Headache in Juvenile Onset Systemic Lupus Erythematosus
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Zülal TATAR, Researcher, Pamukkale University
Other Study IDs: Headache
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2024-12

CONDITIONS: Headache; Juvenile Systemic Lupus Erythematosus
MeSH Terms: conditions — Headache

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of our study was to compare individuals with juvenile onset systemic lupus erythematosus with and without headache in terms of pain, pain catastrophizing behavior, demographic and individual disease-related factors that may affect headache and temporomandibular joint dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with Juvenile Onset Systemic Lupus Erythematosus by the Pediatric Rheumatology Clinic
* Being between the ages of 8-25,
* Having stable symptoms and medications
* Being willing to participate in the study

Exclusion Criteria:

* Patients with neuropsychiatric disorders not associated with Juvenile Onset Systemic Lupus Erythematosus (such as history of epilepsy, electrolyte imbalance, or medication side effects)
* History of headache before juvenile onset systemic lupus erythematosus diagnosis
* Presence of another concomitant rheumatic disease
* Having cognitive impairment to the extent of not being able to cooperate

Ages: 8 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study will include individuals ages 8 to 25 years who are receiving treatment for Juvenile Onset Systemic Lupus Erythematosus at a university hospital in Turkey, and meet the inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2024-10-24 (Actual); Primary Completion 2024-12-24 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
McGill Melzack Pain Questionnaire | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  McGill Melzack Pain Questionnaire consists of four sections. The total score is between 0 and 78 As the score increases, the pain level worsens.
Pain Catastrophizing Scale for Children | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  Pain Catastrophizing Scale for Children is a revised questionnaire consisting of 13 items. Scores range from 0 to 52. Higher score indicate that worse catastrophizing.
Pain Catastrophizing Scale for Parents | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  It consists of 13 items. The scores range from 0 to 52. Higher score indicate that worse catastrophizing.
Fonseca Anamnestic Questionnaire | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  Temporomandibular joint dysfunction was assessed using the Fonseca Anamnestic Questionnaire. The Fonseca Anamnestic Questionnaire consists of 10 questions. The participant is asked to answer each question as 'Yes' (10 points), 'No' (0 points) and 'Sometimes' (5 points). The questionnaire score is scored for all questions and the severity of Temporomandibular joint dysfunction is classified according to the total score. It is classified as no Temporomandibular joint dysfunction (0-15 points), mild Temporomandibular joint dysfunction (20-40 points), moderate Temporomandibular joint dysfunction (45-65 points), severe Temporomandibular joint dysfunction (70-100).
Demographic and disease-related data | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  Such as forehead pain, jaw pain, sore throat, ear pain, neck pain, shoulder pain, psychiatric support, parental togetherness, parents being involved in the child's life, use of vitamin supplements, history of hospitalization due to headache, previous surgery, hearing problems, recurrent sinus infection, recurrent sore throat, asthma, snoring, snoring during sleep, vomiting with headache, reflux, recurrent stomach pain, numbness and tingling with headache, easy bleeding and bruising, eating disorder, frequent nosebleeds, diabetes, obesity, sudden weight loss were recorded as 'yes/no'.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)